CLINICAL TRIAL: NCT07035353
Title: A Clinical Study Evaluating the Efficacy and Safety of Real-world T-DXd in Treating Chinese Patients With HER2 Overexpression and HER2 Underexpression Advanced Breast Cancer
Brief Title: A Real-world Clinical Study of T-DXd for the Treatment of Chinese Patients With HER2 Overexpressing and HER2 Underexpressing Advanced Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDXD2025
Record Dates: First submitted 2025-06-12; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: HER2 Overexpression; Advanced Stage Breast Cancer; Low Expression of HER2
MeSH Terms: interventions — trastuzumab deruxtecan; Isovaleryl-CoA Dehydrogenase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HER2 overexpression in advanced breast cancer patients
  Interventions: Drug: T-DXd (DS8201) 5.4 mg/kg, IVD, 1 cycle every 21 days.
- Patients with advanced breast cancer with low HER2 expression
  Interventions: Drug: T-DXd (DS8201) 5.4 mg/kg, IVD, 1 cycle every 21 days.

INTERVENTIONS:
Drug: T-DXd (DS8201) 5.4 mg/kg, IVD, 1 cycle every 21 days. — The treatment plan will be recommended to the subject by the treating physician in accordance with current clinical practice guidelines and clinical practice, and the patient's decision to receive T-DXd (DS8201) should precede enrollment in this study. The strategy for administering a particular treatment to a subject is not determined a priori by the trial protocol, but should be in accordance with current clinical practice. Because of the non-interventional nature of this study, this study does not alter or interfere with the patient's actual current medical practice.

SUMMARY:
The study is an open, prospective study to collect data on the efficacy and safety of T-DXd (DS8201) in Chinese patients with HER2 overexpressing and HER2 underexpressing advanced breast cancer in actual clinical practice in China.

Cohort A:

HER2 overexpressing patients with advanced breast cancer

Cohort B:

HER2 underexpressing patients with advanced breast cancer A total of 400 subjects will be enrolled in the program, with 200 enrolled in Cohort A and 200 enrolled in Cohort B. The study will be conducted by a physician in accordance with current clinical practice. The treatment plan will be recommended to the subjects by the treating physician based on the current clinical practice guidelines in conjunction with the clinical practice, and the patient's decision to be treated with T-DXd (DS8201) should precede enrollment in this study. Because of the non-interventional nature of this study, this study does not alter or interfere with clinician treatment decisions, and the actual medical practice of patients.

Inclusion in the study after the first treatment with the drug is based on inclusion/exclusion criteria. Subject enrollment in this study should be within 2 months of the subject's first dose of medication and prior to the first efficacy assessment. Demographic data, past medical and treatment history, ECOG score, vital signs + physical examination, laboratory tests, objective tumor evaluation, coadministration/concomitant therapy, adverse events, time to progression/death, and subsequent antitumor therapy were collected at baseline, during treatment, and at subsequent follow-up. Imaging evaluation was performed according to RECIST 1.1 criteria. Adverse events evaluation criteria were based on NCI-CTCAE version 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Must be competent and able to sign and date an Institutional Review Board (IRB) or Ethics Committee (EC)-approved ICF prior to any study-specific procedure or trial.
2. Female patients aged ≥18 years with advanced breast cancer who are adults.
3. Pathologically confirmed breast cancer that meets the following criteria:

   1. unresectable or metastatic, with evidence of recurrent or metastatic disease.
   2. HER2 overexpression, or HER2 hyperexpression as determined by the central laboratory in accordance with the American Society of Clinical Oncology-Society of American Pathologists guidelines.
4. Patients must have measurable lesions according to RECIST 1.1 criteria.
5. Unmenopausal, menopausal, and perimenopausal female patients were allowed to be enrolled.
6. Prior antitumor therapy against recurrent metastatic disease is allowed.

Exclusion Criteria:

1. Early stage breast cancer
2. Patients who do not meet the criteria for HER2 overexpression and HER2 underexpression.
3. Female patients during pregnancy or lactation.
4. Patients deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving T-DXd (DS8201) for HER2 overexpression and HER2 underexpression advanced breast cancer in actual clinical practice in China Chinese patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2035-05-01 (Estimated)

PRIMARY OUTCOMES:
To assess progression-free survival (PFS) of Chinese patients with advanced breast cancer with HER2 overexpression and HER2 underexpression treated with real-world T-DXd (DS8201). | through study completion, an average of 1 year